CLINICAL TRIAL: NCT05356026
Title: The Effect of the Online Postpartum Follow-up on Depression and Postpartum Adaptation: A Randomized Controlled Study
Brief Title: Online Postpartum Follow-up on Depression and Postpartum Adaptation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Şengül Yaman Sözbir, Assoc. Prof., Gazi University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2020/93
Record Dates: First submitted 2022-04-20; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Postpartum Depression; Postpartum Adaptation
Keywords: Postpartum depression; postpartum adaptation; online follow-up; postpartum care; nurse
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online follow up group (Experimental): The women in the experimental group were administered three follow-ups (education/consultancy) in line with the timing and content in the T.R. Ministry of Health Postpartum Care Management Guide (2014). The follow-ups were performed using the Zoom® program, which enabled video talk.
  Interventions: Other: Online postpartum follow-up
- Routine follow up group (No Intervention): The women in the control group received the routine follow-up and care provided by the hospital.

INTERVENTIONS:
Other: Online postpartum follow-up — The women in the experimental group were administered three follow-ups (education/consultancy) in line with the timing and content in the T.R. Ministry of Health Postpartum Care Management Guide (2014). The follow-ups were performed using the Zoom® program, which enabled video talk.
  Arms: Online follow up group

SUMMARY:
Objective: To determine the effect of online postpartum follow-up on depression and postpartum adaptation.

Design: A parallel-randomized-controlled study Setting: During 2021 in Turkey Participants: 52 women in the postpartum period Measurements: Data were collected through the Personal Information Form, the Follow-up Form, the Edinburgh Postpartum Depression Scale (EPDS), and the Postpartum Self-Assessment Scale (PSAS). The women in the experimental group were administered three follow-ups (education/consultancy) in line with the timing and content in the T.R. Ministry of Health Postpartum Care Management Guide (2014). The follow-ups were performed using the Zoom® program, which enabled video talk. The women in the control group received the routine follow-up and care provided by the hospital.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of online postpartum follow-up on depression and postpartum adaptation.

Methods:

Design:

This study utilized a parallel-randomized-controlled experimental design using single-center, stratified randomization (parity: primiparous-multiparous; mode of delivery: vaginal-cesarean).

Participants:

The target population of the study was women in the postpartum period who gave birth in the gynecology service of a university hospital at Ankara (capital city of Turkey) between 10.03.2021 and 20.08.2021. The sample size was determined using power analysis, which included using the information in a similar study conducted before (Serçekuş and Mete, 2010). Analysis was performed using the G power 3.1 version. The minimum number of participants in each group was determined 26, which was 52 in total (α=0,05, 1- β=0,95). However, considering the rate of loss in the source taken as reference (19.7%), a total of 62 individuals were randomized for the sample. In this regard, the participants were planned to be excluded from the study in cases when the mother or the baby is hospitalized, participants want to leave the study, the data collection tools are not filled in, or the participants cannot be reached for education/consultancy. However, no loss of the sample was experienced after the randomization. Post-hoc analysis conducted using the study findings showed that according to the Edinburgh Postpartum Depression Scale mean scores, the power of the study was high (Power [1-β]: 0.99, Effect Size [Cohen's d]: 1.084), and the number of the sample was adequate.

Reliability and Validity of the Study:

Inclusion criteria were determined to prevent selection bias. Hence, the study included volunteer women who were at least literate, who had a live birth, who were aged 18 and over, who were within the first 48 hours of the postpartum period, and who had technical possibilities to use the zoom application.

The women included in the sample were randomized to prevent any bias in distribution. Stratified randomization was performed for the randomization of the study sample. In this regard, the women were divided into 4 stratified groups in terms of parity (primiparous, multiparous) and mode of delivery (vaginal, cesarean).

1. st Stratum Group: Women who were primiparous and had a vaginal delivery
2. nd Stratum Group: Women who were primiparous and had a cesarean section
3. rd Stratum Group: Women who were multiparous and had a vaginal delivery
4. th Stratum Group: Women who were multiparous and had a cesarean section. Women were assigned to the stratified groups using simple randomization. Hence, for each stratum, the first pregnant woman was assigned to the experimental or control group by flipping a coin. The second pregnant woman was assigned to the opposite group. This procedure was repeated as the 3rd, 5th, and 7th, etc. every two pregnant women. Randomization was done by the researcher and no blinding was performed.

Pre-tests were filled in and randomization assignments of the women were performed by an independent nurse to prevent assignment bias. Data obtained from the studies that aimed to prevent reporting bias were coded by an independent researcher as A and B and put in the SPSS program, and data analysis was performed by an independent statistician.

Data Collection:

Data were collected through the Personal Information Form, the Follow-up Form, the Edinburgh Postpartum Depression Scale (EPDS), and the Postpartum Self-Assessment Scale (PSAS).

The Personal Information Form: The form was composed of nine multiple-choice questions that collected data about women's socio-demographic characteristics.

The Follow-up form: This form was conducted to determine problems experienced by women during follow-ups as well as their educational needs. The form prepared in line with the T.R. Ministry of Health Postpartum Care Management Guide (2014) is composed of 25 questions. Participating women were asked open and closed-ended questions that collected data to evaluate their sleep condition, amount and color of bleeding, pain, urinary problems, constipation, psychological condition, domestic violence, breastfeeding, breast problems, personal hygiene, blood incompatibility, exercise, medicine support, benefits of breast milk and things to do to increase it, postpartum family planning, newborn care, and emergency cases that could happen in the postpartum period.

The Edinburgh Postpartum Depression Scale (EPDS): The scale developed by Cox et al. (1987) is utilized to determine the risk of depression in the postpartum period and to measure its level and severity. EPDS is a self-report scale that has one sub-scale and 10items rated on a 4-point Likert scale. The scores to be obtained from the scale range between 0 and 30. Turkish adaptation of the EPDS was performed by Aydın et al. (2004). The cut-off point of the scale is 12, and women who have higher scores than the total cut-off point are considered to be in the risk group. Cronbach's alpha value was found to be 0.72 in the reliability-validity analysis of the scale. In this study, Cronbach's alpha value was found 0.823.

The Postpartum Self-Assessment Scale (PSAS): The Postpartum Self-Assessment Scale was developed by Lederman and Weingarten (1981). The scale aims to assess the adaptation of women in the postpartum period to maternity. Turkish reliability and validity of the scale were performed by Taşçı and Mete (2007). The scale has 82 items rated on a 4-point Likert scale and has seven sub-scales with 10 to 13 items in each. These sub-scales are the quality of the relationship between partners, partners' perception of participation in childcare, gratification with the labor experience, satisfaction with life situations and circumstances, confidence in the ability to cope with the tasks of motherhood, satisfaction with motherhood, and infant care, and support for the maternal role from friends and other family members. The scores to be obtained from the scale range between 82 and 328. Lower scores indicate good compatibility in that area. In the Turkish reliability and validity of the scale, Cronbach's alpha value was found 0.87. This study found Cronbach's alpha coefficient as 0.936.

Intervention Women who gave birth in the gynecology service were met face-to-face within the first 24 hours of the postpartum period, informed about the purpose of the study as well as the implementation process, and those who agreed to participate in the study were identified. Then women who met the research criteria were determined.

Pre-tests (EPDS and PSAS) were administered after these women were asked to sign informed consent forms. After randomization was performed by the chief nurse of the clinic, the women's groups (experimental or control) were identified, and women's contact details were received.

Experimental Group:

The women in the experimental group were administered three follow-ups (education/consultancy) in line with the timing and content in the T.R. Ministry of Health Postpartum Care Management Guide (2014). The follow-ups were performed using the Zoom® program, which enabled video talk.

The problems and education topics in the follow-ups were as follows:

1. st Follow-up: The first follow-up was performed in the 2nd to 5th days of the postpartum period and included the evaluation of the overall condition (sleep, rest, weakness), evaluation of bleeding- lochia, evaluation of urinary problems, evaluation of pain (back, chest, headache, etc.), evaluation of palpitation/shortness of breath, intestinal problems, evaluation of the psychological condition, evaluation of domestic violence, evaluation of maternal and infant relationship, evaluation of breasts/breastfeeding and education (lochia follow-up, perineal care, wound care for those who had a cesarean section, breast milk/breastfeeding, physical activity, emergency cases).
2. nd Follow-up: The second follow-up was performed in the 13th to 17th days and included the evaluation of the overall condition (sleep, rest, weakness), evaluation of bleeding- lochia, evaluation of urinary problems, evaluation of pain (back, chest, headache, etc.), evaluation of palpitation/shortness of breath, evaluation of intestinal problems, evaluation of the psychological condition, evaluation of domestic violence, evaluation of maternal and infant relationship, evaluation of breasts/breastfeeding and education (frequently encountered problems in the newborn, family planning methods).
3. rd Follow-up: The third follow-up was performed in the 30th to 42nd days and included the evaluation of the overall condition (sleep, rest, weakness), evaluation of bleeding- lochia, evaluation of urinary problems, evaluation of pain (back, chest, headache, etc.), evaluation of palpitation/shortness of breath, evaluation of intestinal problems, evaluation of the psychological condition, evaluation of domestic violence, evaluation of maternal and infant relationship, and evaluation of breasts/breastfeeding.

The content of the education and recommendations for the common problems were prepared using the expert views of six professionals in obstetrics and gynecology nursing, and the content validity was calculated using the Davis Technique (Uğurlu and Akgün, 2019). Content validity index of the education content was found 0,89. During the follow-ups, the problems experienced by either the women or the infants were initially investigated, and standardized recommendations were made for these problems. All the women were asked the same questions, but individualized education and consultancy were given for the problematic cases in the answers. Then standardized education prepared was given through the Zoom program online, using a PowerPoint presentation. The participants were asked 5 questions at the end of each education to test the comprehensibility. Unclear parts in the answers were explained again, and the talks took about 40-60 minutes. After the first follow-up, all the women were sent the education booklet and videos (techniques for pumping breastmilk and postpartum exercise) prepared by the researcher through emails. One week after the first follow-up (between the 30th and 42nd days of postpartum), participating women were administered the EPDS and PSAS again. The data collection tools were put in the Google Forms as online questionnaires and sent to the participants.

Control Group The women in the control group received the routine follow-up and care provided by the hospital. The women were sent the EPDS and PSAS between the 30th to 42nd days of postpartum through email and asked to fill them in.

Data Analysis:

Data were analyzed using the IBM SPSS version 24.0 package program. The normality distribution of the data was analyzed using the Shapiro-Wilk test. Whether the groups were homogenous in terms of some socio-demographic and obstetric features was analyzed using t-test in independent groups in numeric variables and chi-square test in categorical variables. EPDS and PSAS total mean scores of the experimental and control groups were compared using t-test in independent groups. Statistical significance was accepted at 0.05 (p<0.05). The effect size was determined by calculating Cohen's d (small-0.2, medium-0.5, and large effect-0.8). The power of the hypotheses was tested based on a minimum 0.80 power level to determine the real effect in experimental studies.

ELIGIBILITY:
Inclusion Criteria:

Women those,

* aged 18 and over
* at least literate
* who have given a live birth
* in the first 48-hour period of the postpartum period
* who have the technical infrastructure to use the online education application (Zoom)

Exclusion Criteria:

Women those,

* illiterate
* those with a high-risk pregnancy diagnosis
* those who do not want to participate

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2021-03-10 (Actual); Primary Completion 2021-08-20 (Actual); Study Completion 2021-09-28 (Actual)

PRIMARY OUTCOMES:
Postpartum depression | 6 weeks (Test 1: first 24 hours of the postpartum period, Test 2: between the 30th and 42nd days of postpartum period)
  The Edinburgh Postpartum Depression Scale (The scale is a self-report scale that has one sub-scale and 10items rated on a 4-point Likert scale. The scores to be obtained from the scale range between 0 and 30. The cut-off point of the scale is 12, and women who have higher scores than the total cut-off point are considered to be in the risk group.)
Postpartum adaptation | 6 weeks (Test 1: first 24 hours of the postpartum period, Test 2: between the 30th and 42nd days of postpartum period)
  The Postpartum Self-Assessment Scale ((The scale aims to assess the adaptation of women in the postpartum period to maternity. The scale has 82 items rated on a 4-point Likert scale and has seven sub-scales with 10 to 13 items in each. These sub-scales are the quality of the relationship between partners, partners' perception of participation in childcare, gratification with the labor experience, satisfaction with life situations and circumstances, confidence in the ability to cope with the tasks of motherhood, satisfaction with motherhood, and infant care, and support for the maternal role from friends and other family members. The scores to be obtained from the scale range between 82 and 328. Lower scores indicate good compatibility in that area.)

CONTACTS AND LOCATIONS:
Locations (1):
- Gazi University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No